CLINICAL TRIAL: NCT00717678
Title: A Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Prograf (Tacrolimus)/MMF and Extended Release (XL) Tacrolimus /MMF in de Novo Kidney Transplant Recipients
Brief Title: A Randomized Study to Assess the Safety and Efficacy of Prograf vs Prograf-XL in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRGXLKTx-0701-TW
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Transplantation; Transplantation Immunology; Host vs Graft Reaction
Keywords: Immunosuppressant; Combination drug therapy; Graft loss; Randomized controlled trial; Open level method
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf-XL + MMF (Experimental)
  Interventions: Drug: Prograf-XL; Drug: MMF
- Prograf + MMF (Active Comparator)
  Interventions: Drug: Prograf; Drug: MMF

INTERVENTIONS:
Drug: Prograf-XL — oral
  Other Names: tacrolimus extended release; FK506XL; MR4
  Arms: Prograf-XL + MMF
Drug: Prograf — oral
  Other Names: tacrolimus; FK506
  Arms: Prograf + MMF
Drug: MMF — oral
  Other Names: Mycophenolate Mofetil

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Prograf extended release(XL) plus MMF with Prograf plus MMF in de novo kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures
* Patient is a recipient of a primary or retransplanted cadaveric or non-HLA-identical living kidney transplant
* Patient must receive first oral dose of randomized study drug within 48 hours of transplant procedure
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment or upon hospitalization

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a kidney
* Patient has received a kidney transplant from a non-heart beating donor
* Patient has received an ABO incompatible donor kidney
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Patient has significant liver disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range of the investigational site
* Patient has an uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives
* Patient is currently taking or has been taking an investigational drug in the 30 days prior to transplant
* Patient is receiving everolimus or enteric coated mycophenolic acid at any time during the study
* Patient has a known hypersensitivity to tacrolimus, mycophenolate mofetil or corticosteroids
* Patient is pregnant or lactating
* Patient is unlikely to comply with the visits scheduled in the protocol
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The patient and graft survival rates at 6 month post-transplant | 6 months

SECONDARY OUTCOMES:
Efficacy failure at 6-month posttransplant. | 6 months
Incidence of biopsy confirmed acute rejection (Banff > 1) at 6 months and 12 months | 6 months and 12 months
1 year patient and graft survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=PRGXLKTx-0701-TW